CLINICAL TRIAL: NCT03581188
Title: A Randomised Controlled Pilot Trial of Patient-led Surveillance Compared to Clinician-led Surveillance in People Treated for Localised Melanoma.
Brief Title: Patient-led Surveillance Compared to Clinician-led Surveillance in People Treated for Localised Melanoma.
Acronym: MEL-SELF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Melanoma and Skin Cancer Trials Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANZMTG 02.17; ACTRN12616001716459 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2018-06-18; First posted 2018-07-10 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-led surveillance (Experimental): Participants receive a mobile dermatoscope that attaches to their smartphone to take photos of skin lesions for teledermatology, instructions on skin self-examination from the ASICA skin checker App, text and email reminders to perform self-examination every 2 months, an educational booklet 'Your guide to early melanoma', and scheduled visits to their clinician as required.
  Interventions: Device: Patient-led surveillance
- Clinician-led surveillance (Active Comparator): Participants receive an educational booklet 'Your guide to early melanoma' and scheduled visits to their clinician as required.
  Interventions: Behavioral: Clinician-led surveillance

INTERVENTIONS:
Device: Patient-led surveillance — Usual care plus reminders, ASICA instructional videos, a mobile dermatoscope, an app that facilitates store-and-forward teledermatology, and fast-tracked unscheduled clinic visits.
  Arms: Patient-led surveillance
Behavioral: Clinician-led surveillance — Usual care (scheduled clinician visits)
  Arms: Clinician-led surveillance

SUMMARY:
The purpose of this pilot study is to evaluate digitally supported skin self-examination compared to usual care in people treated for localised melanoma.

DETAILED DESCRIPTION:
Patients may be eligible to join this study if they are aged 18 years or above, have been treated for stage 0/I/II melanoma and are attending regular melanoma surveillance follow-ups at the Melanoma Institute Australia (MIA), Royal Prince Alfred Hospital (RPAH) or the Newcastle Skin Check Clinic.

People who are found to be eligible and who consent to participate will be randomised (allocated by chance) to the intervention or usual care in a 1:1 ratio. Usual care group will receive an educational booklet on early melanoma and the usual number of routine clinic visits. In addition to usual care, participants allocated to the intervention group will be required to download a skin checker App to their smartphone and will use a mobile dermatoscope to perform total body skin self-examinations every 2 months for 6 months in total. Email and SMS reminders will also be sent every two months to participants in the intervention group. Participants will be documented on how well they are able to perform a self skin examination, their levels of melanoma-related anxiety, the number of skin lesions biopsied or removed, and the costs of follow-up to the participant and to the healthcare system.

Frequent follow-up of localised melanoma is time and resource intensive, and has not shown improved outcomes. This pilot study will provide evidence on which model is best for follow-up care after treatment for localised melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for stage 0/I/II melanoma and are attending regular melanoma follow-up as indicated by scheduled visit within next 12 months in clinic patient booking system and
* Are able to self-examine;
* Have a suitable study partner (spouse, partner, family member, friend);
* Have a smart phone with access to Wifi / email / SMS text messaging;
* Are able to give informed consent ;
* Have sufficient English language skills to read the materials and complete the questionnaires;

Exclusion Criteria:

* Unable to perform self-examination
* No partner or friend to help with self-examination
* Do not have access to a smart phone with Wifi/email/SMS text messaging
* With a known past or current diagnosis of cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katy Bell, A/Prof, Principal Investigator — University of Sydney
Locations (3):
- Australia (3):
  - Newcastle Skin Check, Newcastle, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drabarek D, Ackermann D, Medcalf E, Bell KJL. Acceptability of a Hypothetical Reduction in Routinely Scheduled Clinic Visits Among Patients With History of a Localized Melanoma (MEL-SELF): Pilot Randomized Clinical Trial. JMIR Dermatol. 2023 Jun 26;6:e45865. doi: 10.2196/45865. PMID 37632976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This pilot randomised clinical trial was conducted at 2 specialist-led clinics in metropolitan Sydney, Australia, and a primary care skin cancer clinic managed by general practitioners in metropolitan Newcastle, Australia between November 2018 and January 2020.
Pre-assignment Details: Of the 481 participants screened from November 1, 2018, to May 24, 2019, for eligibility, 125 were ineligible and 30 could not be contacted, leaving 326 participants who were eligible and contacted. Of them, 100 participants were randomized and enrolled in the trial.
Groups:
- Intervention: Patient-led Surveillance: Patient-led surveillance comprised instructional videos on how to perform SSE, reminders to undertake SSE, a mobile dermatoscope that attached to their smartphone, an app that facilitated store-and-forward teledermatology, and fast-tracked unscheduled clinic visits. They received an educational booklet 'Your guide to early melanoma' and scheduled visits to their clinician as required.
- Control: Clinician-led Surveillance: Participants received an educational booklet 'Your guide to early melanoma'and scheduled visits to their clinician as required.
Period: Overall Study
Arm/Group | Intervention: Patient-led Surveillance | Control: Clinician-led Surveillance
Started | 49 | 51
Completed | 30 | 36
Not Completed | 19 | 15
Not completed — Inclusion criteria not met | 3 | 2
Not completed — Lost to Follow-up | 5 | 5
Not completed — Discontinued intervention | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: Patient-led Surveillance | Control: Clinician-led Surveillance | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (12.3) | 59.7 (11.6) | 58.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 27 | 27 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indigenous status: Neither Aboriginal nor Torres Strait Islander | 41 | 33 | 74
  Indigenous status: Unknown | 8 | 18 | 26
No. of melanomas [Count of Participants; unit: Participants]
  1 | 33 | 43 | 76
  2 | 8 | 5 | 13
  3 or more | 8 | 3 | 11
Melanoma substage (highest substage if multiple primary melanomas) [Count of Participants; unit: Participants] — Melanoma stage was classified according to the 8th American Joint Committee on Cancer. Stages range from 0 where the melanoma is confined to the epidermis (melanoma in situ) through to stage IV where the melanoma has spread to distant organs or lymph nodes.
  Participants
    0 | 18 | 18 | 36
    IA | 27 | 22 | 49
    IB | 3 | 6 | 9
    IIA | 0 | 1 | 1
    IIB | 0 | 2 | 2
    III/IV | 0 | 2 | 2
    Unknown | 1 | 0 | 1
Median time elapsed since diagnosis (IQR) [Median (Inter-Quartile Range); unit: years]
  First melanoma diagnosis | 5.5 [0.1 to 41.2] | 5.9 [0.2 to 41.7] | 5.6 [0.1 to 41.7]
  Most recent melanoma diagnosis | 4.3 [0.1 to 41.2] | 5.6 [0.2 to 41.7] | 4.7 [0.1 to 41.7]
Site [Count of Participants; unit: Participants]
  Sydney | 27 | 28 | 55
  Newcastle | 22 | 23 | 45
Main language spoken at home [Count of Participants; unit: Participants]
  English | 43 | 44 | 87
  Other | 6 | 7 | 13
Marital status [Count of Participants; unit: Participants]
  Single, never married | 2 | 2 | 4
  Married | 38 | 33 | 71
  De facto/committed relationship | 3 | 5 | 8
  Separated/divorced | 0 | 1 | 1
  Widowed | 0 | 3 | 3
  Unknown | 6 | 7 | 13
Level of education [Count of Participants; unit: Participants]
  No formal | 0 | 0 | 0
  Primary school | 0 | 1 | 1
  High school diploma/certificate | 11 | 9 | 20
  Vocational diploma/certificate | 9 | 7 | 16
  Bachelor's degree | 11 | 16 | 27
  Postgraduate degree or higher | 12 | 11 | 23
  Unknown | 6 | 7 | 13
Remoteness (based on postal code) [Count of Participants; unit: Participants]
  Metropolitan area/city | 38 | 42 | 80
  Inner regional/rural area | 5 | 2 | 7
  Unknown | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Eligible and Contacted Patients Who Were Randomised Into the Trial
Description: For the primary outcome (composite primary outcome), the percentage was estimated using the number of patients screened who were eligible and contacted as the denominator and the number of patients who were randomised as the numerator.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Patients Who Were Eligible and Contacted: Patients who were screened, eligible and contacted
Arm/Group | Patients Who Were Eligible and Contacted
Number analyzed (Participants) | 326
Participants | 100

2. Secondary Outcome: Adherence to Recommended Total Body Skin Self Examinations Practice: Frequency of Skin Self-examinations.
Description: Adherence to the national guidelines recommendations on skin self-examination frequency was measured via a patient questionnaire asking participants how often they performed a complete self-examination of their skin over the previous 6 months.
Time Frame: Baseline, at 6 months
Population: There were missing data at baseline for 7 (14%) participants in the control group and 6 (12%) in intervention group; and at follow-up for 15 (29%) in the control group and 19 (39%) in intervention group.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Clinician-led Surveillance: Participants received an educational booklet 'Your guide to early melanoma' and scheduled visits to their clinician as required.
Arm/Group | Intervention: Patient-led Surveillance | Control: Clinician-led Surveillance
Number analyzed (Participants) | 49 | 51
Participants
  Baseline: number analyzed (Participants) | 43 | 44
  Baseline: <2 skin self examinations | 13 | 16
  Baseline: ≥2 skin self examinations | 30 | 28
  Follow-up: number analyzed (Participants) | 30 | 36
  Follow-up: <2 skin self examinations | 3 | 10
  Follow-up: ≥2 skin self examinations | 27 | 26
Statistical Analysis 1: Comparison: Intervention: Patient-led Surveillance vs Control: Clinician-led Surveillance; Odds ratios report differences between groups at follow-up; Test type: Superiority; Odds Ratio (OR) = 3.5, 95% CI 2-sided [0.9 to 14]

3. Secondary Outcome: Adherence to Recommended Total Body Skin Self Examinations Practice: Thoroughness of Skin Self-examination
Description: To calculate this variable, the percentage of participants who examined the whole body skin surface during skin self-examination was calculated. Participants were asked if they performed a complete examination of their skin including hard to see areas such as neck/scalp, bottom and feet.
Time Frame: Baseline, 6 months
Population: There were missing data at baseline for 6 (12%) participants in the control group and 5 (10%) in intervention group; and at follow-up for 15 (29%) in the control and 18 (37%) in the intervention group.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Clinician-led Surveilllance: Participants received an educational booklet 'Your guide to early melanoma' and scheduled visits to their clinician as required.
Arm/Group | Intervention: Patient-led Surveillance | Control: Clinician-led Surveilllance
Number analyzed (Participants) | 49 | 51
Participants
  Baseline: number analyzed (Participants) | 44 | 45
  Baseline: No | 36 | 38
  Baseline: Yes | 8 | 7
  Follow-up: number analyzed (Participants) | 31 | 36
  Follow-up: No | 14 | 23
  Follow-up: Yes | 17 | 13
Statistical Analysis 1: Comparison: Intervention: Patient-led Surveillance vs Control: Clinician-led Surveilllance; Test type: Superiority; Odds Ratio (OR) = 2.2, 95% CI 2-sided [0.8 to 5.7]

4. Secondary Outcome: Successful Submission of Dermoscopic Images for Teledermatology (Intervention Group Only)
Description: The number of times images were successfully submitted for teledermatologist review over the six-month intervention period by intervention group participants (count and percentage presented).
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Patient-led Surveillance
Number analyzed (Participants) | 49
Participants
  0 | 23
  1 | 12
  2 | 12
  3 | 2

5. Secondary Outcome: Number of Skin Clinic Visits Attended (Scheduled and Unscheduled)
Description: Total number of clinic visits attended (both scheduled and unscheduled)
Time Frame: During the 12 months after randomisation
Measure: Median (Inter-Quartile Range); unit: Clinic visits
Arm/Group | Intervention: Patient-led Surveillance | Control: Clinician-led Surveillance
Number analyzed (Participants) | 49 | 51
Clinic visits | 2 [0 to 9] | 1 [0 to 6]
Statistical Analysis 1: Comparison: Intervention: Patient-led Surveillance vs Control: Clinician-led Surveillance; Test type: Superiority; Risk Ratio (RR) = 1.5, 95% CI 2-sided [1.1 to 2.1]

6. Secondary Outcome: Number of Skin Lesions Surgically Excised
Description: This outcome has been assessed by conducting a review of medical records such as histopathology reports and doctor's letters. Descriptive statistics such as median with Interquartile Range of total number of skin lesions surgically excised during 12 months after randomisation were calculated.
Time Frame: During the 12 months after randomisation
Measure: Median (Inter-Quartile Range); unit: Skin lesions surgically excised
Arm/Group | Intervention: Patient-led Surveillance | Control: Clinician-led Surveillance
Number analyzed (Participants) | 49 | 51
Skin lesions surgically excised | 1 [0 to 5] | 0 [0 to 10]
Statistical Analysis 1: Comparison: Intervention: Patient-led Surveillance vs Control: Clinician-led Surveillance; Test type: Superiority; Risk Ratio (RR) = 1.1, 95% CI 2-sided [0.6 to 2]

7. Secondary Outcome: New Subsequent Primary or Recurrent Melanoma Diagnoses
Description: This outcome was assessed by conducting a review of medical records at the clinic. Melanoma stage was classified according to the 8th American Joint Committee on Cancer. Stages range from 0 where the melanoma is confined to the epidermis (melanoma in situ) through to stage IV where the melanoma has spread to distant organs or lymph nodes.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Patient-led Surveillance | Control: Clinician-led Surveillance
Number analyzed (Participants) | 49 | 51
Participants
  0 | 6 | 1
  IA | 2 | 1
  IB | 0 | 0
  IIA | 0 | 0
  IIB | 0 | 0
  IIC | 0 | 1
  Total | 8 | 3
Statistical Analysis 1: Comparison: Intervention: Patient-led Surveillance vs Control: Clinician-led Surveillance; For new melanoma diagnoses, we calculated the difference in proportions and confidence intervals using the χ2 method without continuity correction. We included baseline measurement of the outcome in the models as a covariate to estimate between group difference in change from baseline; Test type: Superiority; Risk Difference (RD) = 10, 95% CI 2-sided [-2 to 23]

8. Secondary Outcome: New Melanoma Diagnoses Prompted by Visit Type
Description: New melanoma diagnoses prompted by visit type such as unscheduled visits and scheduled visits were calculated.
Time Frame: During 12 months after randomisation
Population: During the trial, 11 participants were diagnosed with a subsequent new primary melanoma or recurrence, including 8 in the intervention group and 3 in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Patient-led Surveillance | Control: Clinician-led Surveillance
Number analyzed (Participants) | 49 | 51
Participants
  New melanoma diagnoses at an unscheduled visit | 5 | 0
  New melanoma diagnoses at a scheduled visit | 3 | 3
Statistical Analysis 1: Comparison: Intervention: Patient-led Surveillance vs Control: Clinician-led Surveillance; New melanoma diagnoses prompted at unscheduled visit; Test type: Superiority; Risk Difference (RD) = 10, 95% CI 2-sided [2 to 19]
Statistical Analysis 2: Comparison: Intervention: Patient-led Surveillance vs Control: Clinician-led Surveillance; New melanoma diagnoses prompted at scheduled visit; Test type: Superiority; Risk Ratio (RR) = 0, 95% CI 2-sided [-9 to 10]

9. Secondary Outcome: General Anxiety, Stress, and Depression Measured Using the Depression Anxiety Stress Scales-21
Description: This outcome has been measured using the short version of the Depression Anxiety and Stress Scales (DASS-21). The DASS-21 is a set of three 7-item self-report scales designed to measure the emotional states of depression, anxiety and stress. The depression scale measures dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia and inertia. The anxiety scale measures autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale assesses difficulty relaxing, nervous arousal, and feeling irritable and impatient. Each scale ranges from "Did not apply to me" (0) to "Applied to me very much or most of the time" (3). A higher value is considered a worse outcome.
Time Frame: Baseline, 6 months
Population: There was missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: Clinician-led Surveillance: Participants will receive an educational booklet 'Your guide to early melanoma'and scheduled visits to their clinician as required.
Arm/Group | Intervention: Patient-led Surveillance | Control: Clinician-led Surveillance
Number analyzed (Participants) | 49 | 51
score on a scale
  Baseline: number analyzed (Participants) | 30 | 35
  Baseline | 9.4 (11.2) | 14 (15.3)
  Follow-up: number analyzed (Participants) | 30 | 35
  Follow-up | 6.5 (7.1) | 9.9 (14.5)
Statistical Analysis 1: Comparison: Intervention: Patient-led Surveillance vs Control: Clinician-led Surveillance; Test type: Superiority; Mean Difference (Net) = -1.4, 95% CI 2-sided [-5.8 to 3]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Self-examination of the Skin: Participants will perform self-surveillance of the skin using a dermatoscope device. They will receive guidance from the ASICA skin checker and receive reminders every 2 months to perform self-examination. They will receive an educational booklet 'Your guide to early melanoma' and scheduled visits to their clinician as required.
  Self-examination of the skin: Participants will use a dermatoscope device to conduct self-examination of the skin.
- Control: Participants will receive an educational booklet 'Your guide to early melanoma'and scheduled visits to their clinician as required.
Arm/Group | Self-examination of the Skin | Control
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 1/49 | 0/51
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-examination of the Skin (N=49) | Control (N=51)
Anxiety and confusion arising due to technical difficulties (Psychiatric disorders) | 1 (1) | 0 (0) — One person in the intervention group withdrew due to anxiety and confusion arising due to technical difficulties

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03581188/Prot_SAP_000.pdf